CLINICAL TRIAL: NCT00987532
Title: A Participatory Parental Intervention Promoting Physical Activity in Preschools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Collaborators: Baden-Württemberg Stiftung gGmbH (Other)
Responsible Party: Principal Investigator, Joachim E. Fischer, MD MSc, Director, Mannheim Institute of Public Health, Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MIPH_KITA2008
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Obesity; Physical Activity
Keywords: preschool; participatory intervention; cluster-randomization; children; obesity prevention
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- parent intervention plus gym lessons (Experimental): Parent-focused participatory preschool intervention in addition to twice weekly gym lessons over 6 months. The participatory intervention includes parents, teachers and children.
  Interventions: Behavioral: parent-focused intervention; Behavioral: twice weekly gym lessons
- gym lessons only (Active Comparator): Twice weekly one-hour gym lessons delivered by a specially trained external physical education teacher over 6 months
  Interventions: Behavioral: twice weekly gym lessons

INTERVENTIONS:
Behavioral: parent-focused intervention — The core of the parent-focused intervention is a menu of 15 easy to realize project ideas to promote the everyday physical activity of children and families. The 15 ideas are presented to the parents and teachers via a webpage, a printed book and a film. During a face-to-face meeting, parents and teachers are guided into discussions of their own preschool environment's and community's physical activity shortcomings and encouraged to generate their own ideas of how to enhance the physical activity of their families and preschools. Over the course of three structured follow-up meetings, parents and teachers are instructed to choose maximally 3 to 4 ideas from either the menu or the network's own ideas, and then are empowered to realize and implement them together.
  Other Names: Ene mene fit - Eltern machen mit
  Arms: parent intervention plus gym lessons
Behavioral: twice weekly gym lessons — twice weekly one-hour gym lessons delivered by a specially trained external physical education teacher over 6 months
  Other Names: child-centered physical activity intervention

SUMMARY:
The aim of this study is to test whether a parent-focused participatory intervention in addition to gym lessons can enhance preschoolers physical activity compared to gym lessons alone.

DETAILED DESCRIPTION:
Over the last 20 years, physical activity (PA) in children has rapidly decreased in both developed and developing nations. More effective interventions to prevent inactivity in childhood thus are urgently needed. The preschool years, including the adiposity rebound period, might represent a good window of opportunity. Study literature suggests that targeting parents is crucial for lasting changes in young childrens' behavior. However, it is not known which methods are effective for involving parents in physical activity promotion. Consistent with experience from community-based participatory research, encouraging parents to participate the intervention in terms of content and structure might lead to higher intervention effectivity and sustainability. In our study, we therefore "enriched" a child-centered physical activity intervention in preschools (twice weekly gym lessons over 6 months) with a parent-focused participatory community intervention component.

ELIGIBILITY:
Inclusion Criteria:

* age 3-6 years

Exclusion Criteria:

* severe atopic dermatitis,
* serious acute infectious diseases,
* physical malformations, and
* severe physical disabilities.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1047 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Absolute change in mean accelerometry counts over 6 days | baseline, end of intervention, six months after end of intervention

SECONDARY OUTCOMES:
Body Mass Index | baseline, end of intervention, six months after end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Joachim E. Fischer, MD, M.Sc., Principal Investigator — Mannheim Institute of Public Health, Medical Faculty Mannheim, Heidelberg University
Locations (1):
- Mannheim Institute of Public Health, Medical Faculty Mannheim, Heidelberg University, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] De Bock F, Genser B, Raat H, Fischer JE, Renz-Polster H. A participatory physical activity intervention in preschools: a cluster randomized controlled trial. Am J Prev Med. 2013 Jul;45(1):64-74. doi: 10.1016/j.amepre.2013.01.032. PMID 23790990
- [Derived] De Bock F, Fischer JE, Hoffmann K, Renz-Polster H. A participatory parent-focused intervention promoting physical activity in preschools: design of a cluster-randomized trial. BMC Public Health. 2010 Jan 31;10:49. doi: 10.1186/1471-2458-10-49. PMID 20113522
- See also: webpage of the participatory parent-focused intervention — http://www.ene-mene-fit.de